CLINICAL TRIAL: NCT04001517
Title: A Double-Blind, Placebo-Controlled 16-Week Study of the Cognitive Effects of Oral p38 Alpha Kinase Inhibitor Neflamapimod in Dementia With Lewy Bodies (DLB)
Brief Title: Cognitive Effects of Oral p38 Alpha Kinase Inhibitor Neflamapimod in Dementia With Lewy Bodies
Acronym: AscenD-LB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EIP Pharma Inc (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP19-NFD-501
Record Dates: First submitted 2019-06-07; First posted 2019-06-28 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Dementia With Lewy Bodies (DLB)
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neflamapimod (Experimental): 40 mg capsules administered orally, BID or TID with food for 16 weeks; subjects will follow the BID regimen if weighing <80 kg or the TID regimen if weighing ≥80 kg
  Interventions: Drug: Neflamapimod
- Placebo (Placebo Comparator): 40 mg matching placebo capsules administered orally, BID or TID with food for 16 weeks; subjects will follow the BID regimen if weighing <80 kg or the TID regimen if weighing ≥80 kg
  Interventions: Drug: Neflamapimod

INTERVENTIONS:
Drug: Neflamapimod — Double-Blind, Placebo-Controlled

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, proof-of-principle study of neflamapimod versus matching placebo (randomized 1:1) administered with food for 16 weeks in subjects with DLB. The primary objective is to evaluate the effect of neflamapimod on cognitive function as assessed in a study-specific Cogstate Neuropsychological Test Battery (NTB). Secondary endpoints include the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB), Mini-Mental State Examination (MMSE), Neuropsychiatric Inventory (NPI-10), Timed Up and Go Test, and electroencephalogram (EEG) as a potential biomarker for DLB.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥55 years.
2. Subject or subject's legally authorized representative is willing and able to provide written informed consent.
3. Probable DLB and identified cognitive deficits, according to current consensus criteria (McKeith et al, 2017), specifically one core clinical feature and a positive DaTscan. If a negative DaTscan, but the subject has historical PSG-verified RBD, the subject would also qualify.
4. MMSE score of 15-28, inclusive, during Screening.
5. Currently receiving cholinesterase inhibitor therapy, having received such therapy for greater than 3 months and on a stable dose for at least 6 weeks at the time of randomization. Except for reducing the dose for tolerability reasons, the dose of cholinesterase inhibitor may not be modified during the study.
6. Normal or corrected eye sight and auditory abilities, sufficient to perform all aspects of the cognitive and functional assessments.
7. No history of learning difficulties that may interfere with their ability to complete the cognitive tests.
8. Must have reliable informant or caregiver.

Exclusion Criteria:

1. Diagnosis of any other ongoing central nervous system (CNS) condition other than DLB, including, but not limited to, post-stroke dementia, vascular dementia, Alzheimer's disease (AD), or Parkinson's disease (PD).
2. Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the C-SSRS, or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
3. Ongoing major and active psychiatric disorder and/or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
4. Diagnosis of alcohol or drug abuse within the previous 2 years.
5. Poorly controlled clinically significant medical illness, such as hypertension (blood pressure >180 mmHg systolic or 100 mmHg diastolic); myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would interfere with assessment of drug safety.
6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN), total bilirubin >1.5 × ULN, and/or International Normalized Ratio (INR) >1.5.
7. Known human immunodeficiency virus, hepatitis B, or active hepatitis C virus infection.
8. Participated in a study of an investigational drug less than 3 months or 5 half-lives of an investigational drug, whichever is longer, before enrollment in this study.
9. History of previous neurosurgery to the brain.
10. If male with female partner(s) of child-bearing potential, unwilling or unable to adhere to contraception requirements specified in the protocol.
11. If female who has not has not reached menopause >1 year previously or has not had a hysterectomy or bilateral oophorectomy/salpingo-oophorectomy, has a positive pregnancy test result during Screening and/or is unwilling or unable to adhere to the contraception requirements specified in the protocol.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Alam, MD, Study Director — EIP Pharma
Locations (24):
- United States (22):
  - University of California San Diego (UCSD), La Jolla, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Elite Clinical Research, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic - Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Summit Research Network, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - University of Washington, Seattle, Washington
  - Inland Northwest Research, Spokane, Washington
- Netherlands (2):
  - Brain Research Center, 's-Hertogenbosch
  - Brain Research Center, Amsterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alam JJ, Maruff P, Doctrow SR, Chu HM, Conway J, Gomperts SN, Teunissen C. Association of Plasma Phosphorylated Tau With the Response to Neflamapimod Treatment in Patients With Dementia With Lewy Bodies. Neurology. 2023 Oct 24;101(17):e1708-e1717. doi: 10.1212/WNL.0000000000207755. Epub 2023 Sep 1. PMID 37657939
- [Derived] Jiang Y, Alam JJ, Gomperts SN, Maruff P, Lemstra AW, Germann UA, Stavrides PH, Darji S, Malampati S, Peddy J, Bleiwas C, Pawlik M, Pensalfini A, Yang DS, Subbanna S, Basavarajappa BS, Smiley JF, Gardner A, Blackburn K, Chu HM, Prins ND, Teunissen CE, Harrison JE, Scheltens P, Nixon RA. Preclinical and randomized clinical evaluation of the p38alpha kinase inhibitor neflamapimod for basal forebrain cholinergic degeneration. Nat Commun. 2022 Sep 21;13(1):5308. doi: 10.1038/s41467-022-32944-3. PMID 36130946

RESULTS

PARTICIPANT FLOW:
Groups:
- Neflamapimod TID: 40 mg capsules administered orally TID with food for 16 weeks; subjects followed the TID regimen if Screening weight was ≥80 kg
- Neflamapimod BID: 40 mg capsules administered orally BID with food for 16 weeks; subjects followed the BID regimen if Screening weight was <80 kg
- Placebo TID: 40 mg matching placebo capsules administered orally TID with food for 16 weeks; subjects followed the TID regimen if Screening weight was ≥80 kg
- Placebo BID: 40 mg matching placebo capsules administered orally BID with food for 16 weeks; subjects followed the BID regimen if Screening weight was <80 kg
Period: Overall Study
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo TID | Placebo BID
Started | 20 | 26 | 27 | 18
Completed | 20 | 20 | 26 | 15
Not Completed | 0 | 6 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo capsules matched to neflamapimod capsules, administered orally BID or TID with food for 16 weeks; subjects followed the TID regimen if Screening weight was ≥80 kg or the BID regiment if Screening weight was <80 kg
- Total: Total of all reporting groups
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo | Total
Number analyzed (Participants) | 20 | 26 | 45 | 91
Age, Categorical [Count of Participants; unit: Participants] — Participants were categorized by age (in years), including number of participants and percentage of participants per category. Age was captured at Screening.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 2 | 7 | 11
    >=65 years | 18 | 24 | 38 | 80
Age, Continuous [Mean (Full Range); unit: years] — The full age range of participants as well as the mean age (in years), are provided. Age was captured at Screening.
  years | 72.2 [59 to 84] | 74.5 [63 to 85] | 72.1 [62 to 87] | 72.8 [59 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — The sex/gender of participants were grouped by female and male. Gender was captured at Screening.
  Participants
    Female | 1 | 7 | 6 | 14
    Male | 19 | 19 | 39 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants were categorized by ethnicity. Ethnicity was captured at Screening.
  Participants
    Hispanic or Latino | 0 | 4 | 3 | 7
    Not Hispanic or Latino | 20 | 22 | 42 | 84
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants were categorized by race. Race was captured at Screening.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 1 | 1
    White | 20 | 26 | 44 | 90
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participants were grouped by country of participation. Country was determined based on site where participant was enrolled.
  participants
    Netherlands | 3 | 4 | 6 | 13
    United States | 17 | 22 | 39 | 78
MMSE [Mean (Standard Deviation); unit: units on a scale (range 0-30)] — Participant's Screening Mini-Mental State Examination (MMSE) mean score and standard deviation is provided. MMSE evaluates orientation, memory, concentration, language and praxis. Scores range from 0 to 30 with lower scores indicating greater cognitive impairment.
  units on a scale (range 0-30) | 23.6 (3.7) | 22.4 (3.7) | 23.0 (4.1) | 23.0 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Composite Z-score of a Study-specific Neuropsychological Test Battery (NTB) Including Tests From Cogstate Battery, Letter Fluency Test and Category Fluency Test
Description: Change from Baseline to Week 4, Week 8, and Week 16 in the composite z-score of a study-specific Neuropsychological Test Battery (NTB) that included the following six tests: Cogstate Detection test (DET), Cogstate Identification test (IDN), Cogstate One Card Learning test (OCL), Cogstate One Back test (ONB), Letter Fluency Test, and Category Fluency Test (CFT). Each score on the individual tests was converted to a z-score, and then a total z-score for the composite was calculated, in which each test is weighted equally. As the analysis is based on z-scores, there is no minimum or maximum value. A z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A positive change in z-score indicate an improvement in cognition, i.e., a better outcome; and a negative change in z-score indicates a worsening in cognition, i.e., a worse outcome.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, all time points at which NTB was assessed utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All subjects with a baseline and at least one on-treatment NTB evaluation. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Z-Score
Groups:
- Placebo: 40 mg matching placebo capsules administered orally TID or BID with food for 16 weeks; subjects followed the TID regimen if Screening weight was ≥80 kg and the BID regimen if Screening weight was <80 kg
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
Number analyzed (Participants) | 19 | 20 | 37
Z-Score
  Baseline | 0.06 (0.17) | 0.02 (0.15) | 0.05 (0.11)
  Week 4 | 0.17 (0.14) | -0.08 (0.18) | -0.05 (0.13)
  Week 8 | 0.28 (0.16) | -0.12 (0.18) | 0.05 (0.17)
  Week 16 | 0.21 (0.18) | -0.08 (0.21) | -0.03 (0.14)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Placebo; This was an exploratory trial and no explicit a priori hypothesis was established and contained in the protocol. As such, no formal power calculations were conducted. The primary objective of the study was to evaluate the effects of neflamapimod on cognition, and accordingly the primary endpoint was change in combined z-score of the six tests in the NTB, analyzed by Linear Mixed Effects (LME) model for repeated measures; Test type: Superiority; p = 0.049, Mixed Models Analysis — The comparison is of neflamapimod 40mg TID to placebo. The p-value was not adjusted for multiple comparisons; Mean Difference (Net) = 0.175, 95% CI 2-sided [0.001 to 0.345] — The comparison is of neflamapimod 40mg TID to placebo. The positive value represents a better outcome with neflamapimod 40mg treatment vs. placebo
Statistical Analysis 2: Comparison: Neflamapimod TID vs Neflamapimod BID vs Placebo; Test type: Superiority — Comparison of combined neflamapimod groups vs. placebo; p > 0.2, Mixed Models Analysis

2. Secondary Outcome: Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB)
Description: Change in Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) score from Baseline to Week 8 and Week 16 based on semi-quantitative scoring of six domains (i.e., "box": 1) memory, 2) orientation, 3) judgement & reasoning, 4) home & hobbies, 5) community affairs, and 6) personal care. The CDR score ranges from 0 (no impairment), 0.5 (questionable impairment), 1 (mild impairment), 2 (moderate impairment), and 3 (severe impairment). The domain (box) scores are then added for a Sum of Boxes score. With six domains, the CDR-SB score then ranges from 0 to 18; with higher scores indicated worse outcomes.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, both time points at which CDR-SB was assessed (week 8 and 16) was utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All subjects with a baseline and at least one on-treatment CDR-SB evaluation. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
Number analyzed (Participants) | 20 | 20 | 37
Scores on a scale
  Week 8 | 0.11 (0.2) | 0.19 (0.3) | 0.76 (0.25)
  Week 16 | 0.34 (0.2) | 0.34 (0.18) | 0.86 (0.32)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Placebo; Test type: Superiority — Comparison of combined neflamapimod 40mg TID vs. placebo. The p-value is not adjusted for multiple comparisons; p = 0.007, Mixed Models Analysis — Comparison of combined neflamapimod dose groups vs. placebo utilizing mixed model for repeated measures with baseline as a covariate. The p-value is not adjusted for multiple comparisons; Mean Difference (Net) = -0.56, 95% CI 2-sided [-0.96 to -0.16] — The comparison is of neflamapimod 40mg TID to placebo. A negative value indicates improvement compared to placebo
Statistical Analysis 2: Comparison: Neflamapimod TID vs Neflamapimod BID vs Placebo; A secondary analysis was conducted comparing the combined neflamapimod dose groups vs. placebo; Test type: Superiority; p = 0.023, Mixed Models Analysis — Mixed model for repeated measures with baseline as a covariate. The p-value was not adjusted for multiple comparisons; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.83 to -0.06] — Comparison of combined neflamapimod dose groups vs. placebo. Negative values represents a better outcome with neflamapimod relative to placebo

3. Secondary Outcome: Mini-Mental State Examination (MMSE)
Description: The Mini-Mental State Examination (MMSE) is a general measure of cognition that assesses orientation, memory, concentration, language, and praxis. Scores range from 0 to 30 with lower scores indicating greater cognitive impairment, i.e. a worse outcome). The MMSE was assessed at Week 8 and Week 16 during the study.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, both time points at which MMSE was assessed (week 8 and 16) was utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All subjects with a baseline and at least one on-treatment MMSE evaluation. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
Number analyzed (Participants) | 20 | 21 | 37
Scores on a scale
  Week 8 | 0.11 (0.74) | 0.08 (0.64) | -0.59 (0.38)
  Week 16 | -0.85 (.49) | -1.75 (0.67) | -0.53 (0.49)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Neflamapimod BID vs Placebo; Test type: Superiority; p > 0.2, Mixed Models Analysis

4. Secondary Outcome: Neuropsychiatric Inventory (NPI-10) - Mean Change in Hallucinations Domain Score
Description: The NPI-10 consists evaluates ten domains: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor activity. If caregiver reports symptoms within a domain then the caregiver rates the frequency of the symptoms on a 4-point scale, and severity on a 3-point scale. Total score for each domain is the frequency score multiplied by the severity score; i.e. the domain score (e.g. for hallucinations) for any one domain ranges from 0-12, with higher scores indicating worsening. A secondary objective of this study was to evaluate the effect of neflamapimod in four specific domains, specifically depression (dysphoria), anxiety, hallucinations, and agitation/aggression, in neflamapimod-treated subjects compared to placebo-recipients. Of these four, the only domain in which more than one-quarter of the patients reported symptoms is hallucinations, and the result of this analysis is reported.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, all time points at which NPI-10 was assessed (weeks 4, 8 and 16) was utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All subjects with a baseline and at least one on-treatment NPI-10 evaluation. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Neflamapimod 40 mg BID: 40 mg capsules administered orally BID with food for 16 weeks; subjects followed the BID regimen if Screening weight was <80 kg
Arm/Group | Neflamapimod 40 mg BID | Neflamapimod TID | Placebo
Number analyzed (Participants) | 9 | 8 | 10
Score on a scale
  Week 4 | 0.1 (.875) | -1.71 (1.23) | 0.56 (0.697)
  Week 8 | 0.63 (.46) | -0.86 (1.22) | 0.86 (0.61)
  Week 16 | 3.29 (1.97) | -0.5 (1.2) | 1.71 (1.19)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Placebo; Test type: Other; p = 0.15, Mixed Models Analysis; Mean Difference (Net) = -1.53, 95% CI 2-sided [-3.61 to .55]
Statistical Analysis 2: Comparison: Neflamapimod 40 mg BID vs Neflamapimod TID vs Placebo; Comparison of combined neflamapimod groups (i.e., all neflamapimod) vs. placebo; Test type: Superiority; p = 0.077, Mixed Models Analysis; Mean Difference (Net) = -1.31, 95% CI 2-sided [-5.03 to 2.34]

5. Secondary Outcome: International Shopping List Test (ISLT) - Immediate Recall
Description: The International Shopping List Test (ISLT) was developed specifically to assess verbal list learning and memory in people from different language and cultural backgrounds. 12 words, consisting to items typically in a grocery shopping list in the specific culture are provided verbally, and subject asked to recall ask many words as possible. The immediate recall score consists of the number of words that the subject correctly repeats during three consecutive trials immediately following provision of words. The range is then from 0 to 36 (12 words maximum in each of 3 trials), with higher scores (i.e., the more words recalled) reflecting better outcomes.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, both time points at which ISLT was assessed (Weeks 4, 8 and 16) was utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All participants with at least one on-treatment ISLT immediate recall evaluation available. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
Number analyzed (Participants) | 20 | 20 | 41
Scores on a scale
  Change from baseline to week 4: number analyzed (Participants) | 17 | 20 | 41
  Change from baseline to week 4 | 0.29 (1.08) | -1.24 (0.61) | 0.11 (0.54)
  Change from baseline to week 8: number analyzed (Participants) | 9 | 12 | 29
  Change from baseline to week 8 | 2.11 (1.66) | -0.75 (1.37) | 0.41 (0.65)
  Change from baseline to week 16 | 0.30 (1.04) | 0.11 (.99) | -0.15 (.46)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Neflamapimod BID vs Placebo; Test type: Superiority; p > 0.2, Mixed Models Analysis; Mean Difference (Net) = 0.32, 95% CI 2-sided [-1.27 to 1.91] — Comparison of change from baseline over course of study for NFMD 40mg TID vs. placebo

6. Secondary Outcome: Timed Up and Go Test (TUG)
Description: The Timed Up and Go test assesses function mobility, and was included in the study to evaluate the effects of neflamapimod on motor function. The TUG measures the time in seconds that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. The TUG was evaluated at Baseline, and Weeks 8 and 16 of the study. There is no minimum or maximum value for this test, though in Parkinson's disease patients values above 11.5 seconds was associated with an increased risk of falls and each one second increase in the time required to complete the TUG is associated with a 5.4% increase in the risk of falls (Arch Phys Med Rehabil. 2013;94: 1300-1305). That is, an increase in the time required to complete the TUG is a worse outcome.
Time Frame: As the analysis was by Mixed Model for Repeated Measures, both time points at which the TUG was assessed (week 8 and 16) was utilized in the analysis. The difference reported is the mean difference over the entire course of the study.
Population: All subjects with a baseline and at least one on-treatment TUG evaluation. As placebo given twice or three times a day would not be expected to differences in outcome, per the protocol and statistical analysis plan (SAP) the placebo group was considered as one group, regardless of whether they received placebo BID or TID.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
Number analyzed (Participants) | 20 | 20 | 37
Seconds
  Week 8 | -0.2 (0.5) | 1.0 (0.9) | 0.4 (0.4)
  Week 16 | -1.4 (1.0) | 1.3 (0.7) | 1.5 (0.9)
Statistical Analysis 1: Comparison: Neflamapimod TID vs Placebo; Test type: Other; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = -1.4, 95% CI 2-sided [-2.6 to -0.2] — Mean difference for the comparison of 40 mg TID vs. placebo is reported
Statistical Analysis 2: Comparison: Neflamapimod TID vs Neflamapimod BID vs Placebo; Test type: Superiority — Comparison of combined neflamapimod dose groups vs. placebo; p = 0.044, Mixed Models Analysis; Mean Difference (Net) = -1.36, 95% CI 2-sided [-2.69 to -0.04]

7. Secondary Outcome: Quantitative Electroencephalogram (qEEG)m - Dominant Peak Frequency Over Parietal Lobe
Description: Change in quantitative electroencephalogram (qEEG) parameters with the subject awake in accordance with the 10-20 International System of Electrode placement was to be evaluated as a potential biomarker for DLB. However, due to COVID19 related restrictions, baseline and week 16 EEG recordings were obtained only in limited number of subjects. As slowing of the dominant frequency band by qEEG over posterior aspects of the brain has been recognized to be prominent in DLB, the change in the dominant frequency band over the parietal lobe in Hz from baseline to week 16 is reported. This is a continuous variable with no minimum or maximum. A decrease in the frequency (i.e., slowing) reflects worsening of disease, while a positive treatment effect would be an increase in the frequency. With the limited number of subjects formal statistical analysis was not conducted.
Time Frame: 16 weeks
Population: All subjects with a baseline and week 16 EEG recording.
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Neflamapimod TID | Placebo
Number analyzed (Participants) | 6 | 12
Hz | 0.24 (1.06) | 0.36 (0.95)

ADVERSE EVENTS:
Time Frame: AEs occurring from when the subject signed the ICF until the last study event were collected. (Study Duration = 16 weeks) Any AEs occurring before the start of treatment (i.e., before the first dose of the investigational product) were recorded in the medical history.
Arm/Group | Neflamapimod TID | Neflamapimod BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/26 | 2/45
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/26 | 4/45
Other Adverse Events (participants affected / at risk) | 8/20 | 8/26 | 17/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neflamapimod TID (N=20) | Neflamapimod BID (N=26) | Placebo (N=45)
New brain lesions of unclear etiology (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diagnosis of brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intraparenchymal hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Internal bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neflamapimod TID (N=20) | Neflamapimod BID (N=26) | Placebo (N=45)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 4 (5)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04001517/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT04001517/SAP_001.pdf